CLINICAL TRIAL: NCT01206114
Title: Evaluation of the Effectiveness of Vaccination With 2009 H1N1 Vaccines During Influenza Season 2010-11
Status: Completed | Type: Observational
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Responsible Party: Sponsor
Other Study IDs: H1N1-495-10THL; 2010-021033-30 (EudraCT Number); R10075M (Other: The ethics committee of the Pirkanmaa Hospital District (PSHP)); 81/2010 (Other: Finnish Medicines Agency)
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Influenza Caused by the 2009 H1N1 Influenza Virus
Keywords: 2009 H1N1 influenza; vaccination; pandemic; effectiveness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — nasal/oral swabs, serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vaccinated persons: The participants have taken one or more doses of 2009 H1N1 vaccine, either as a monovalent vaccine or as a part of a trivalent seasonal 2010-2011 influenza vaccine
  Interventions: Other: Follow-up
- Not (yet) vaccinated persons: The participants do not want to take any 2009 H1N1 vaccine or have not received any yet
  Interventions: Other: Follow-up

INTERVENTIONS:
Other: Follow-up — Questionnaires, interviews, nasal/oral and serum samples, register data
  Groups: Vaccinated persons
Other: Follow-up — Questionnaires, interviews, nasal/oral and serum samples, register data
  Groups: Not (yet) vaccinated persons

SUMMARY:
A cohort of 3000 adults is followed to evaluate the effectiveness of the monovalent 2009 H1N1 vaccines used 2009-2010 and seasonal influenza vaccines used 2010-2011 in preventing the first laboratory-confirmed 2009 H1N1 influenza during the influenza season 2010-11.

DETAILED DESCRIPTION:
In the beginning of the study, changes in the background information collected in the original study (conducted 2009-2010) are asked with a questionnaire. Information on influenza vaccinations is collected with vaccination cards and monthly short message service (SMS), and verified in registers, if needed. If an epidemic caused by the 2009 H1N1 virus starts in Finland, the participants are asked to actively report symptoms of influenza like illnesses (ILI). The symptoms are also monitored by weekly SMS. In case of ILI, nasal and oral swabs are collected to verify the 2009 H1N1 influenza cases. Paired serum samples are collected at the acute on convalescence phase of the disease. The occurrence of laboratory-confirmed 2009 H1N1 influenza cases is compared between vaccinated and not (yet) vaccinated persons.

ELIGIBILITY:
Inclusion criteria for the interview follow-up:

* Participating in the study "Evaluation of a vaccination campaign with A(H1N1)v pandemic vaccines: a prospective cohort study" (AH1N1-483-09THL)
* Assigned to use the services of Tampere health care centre;
* Written consent for the interview follow-up phase obtained by mail;
* Able to adhere to all protocol-required study procedures without any special burden or risk, as judged by the participant himself/herself

Inclusion criteria for the confirmation of 2009 H1N1 influenza cases:

* Participating in the study interview follow-up of the current study 'Evaluation the effectiveness of vaccination with 2009 H1N1 vaccines during influenza season 2010-11 (H1N1-495-10THL)
* Assigned to use the services of Tampere health care centre
* Written informed consent for the confirmation phase obtained at the first study visit
* Able to adhere to all protocol required study procedures without any special burden or risk, as judged by the investigator or designate

Exclusion criteria:

* No specific exclusion criteria will be applied

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participation in the study will be offered to all participants of the cohort study "Evaluation of a vaccination campaign with A(H1N1)v pandemic vaccines: a prospective cohort study" AH1N1-483-09THL, who still live in the study area (city of Tampere) and who have complied to the SMS or phone follow-up. The eligibility criteria of the original study AH1N1-483-09THL were: full legal competence; community-dwelling; age 18 to 75 years, written informed consent obtained; able to communicate fluently in Finnish or Swedish and able to adhere to all protocol required study procedures without any special burden or risk. Originally, 3500 persons participated in the study
Sampling Method: Non-Probability Sample
Enrollment: 2351 (Actual)
Dates: Start 2010-09; Primary Completion 2011-04 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
To determine the effectiveness of 2009 H1N1 influenza vaccination in preventing the first episode of laboratory-confirmed influenza caused by the 2009 H1N1 virus during the season 2010-11 among vaccinated adults as compared to unvaccinated adults | September 2010 to April 2011

SECONDARY OUTCOMES:
To explore the ability of different vaccination regimens to prevent 2009 H1N1 influenza | September 2010 to April 2011
To explore the effectiveness of the 2009 H1N1 vaccines in subgroups stratified by age | September 2010 to April 2011
To evaluate the incidence, severity and possible complications of laboratory-confirmed infection with the 2009 H1N1 influenza virus | September 2010 to April 2011

CONTACTS AND LOCATIONS:
Overall Officials: Terhi M Kilpi, MD, PhD, Principal Investigator — Finnish Institute for Health and Welfare
Locations (1):
- National Institute for Health and Welfare, Tampere, Finland

REFERENCES:
- [Derived] Syrjanen RK, Jokinen J, Ziegler T, Sundman J, Lahdenkari M, Julkunen I, Kilpi TM. Effectiveness of pandemic and seasonal influenza vaccines in preventing laboratory-confirmed influenza in adults: a clinical cohort study during epidemic seasons 2009-2010 and 2010-2011 in Finland. PLoS One. 2014 Sep 29;9(9):e108538. doi: 10.1371/journal.pone.0108538. eCollection 2014. PMID 25265186